CLINICAL TRIAL: NCT01793961
Title: Effects of Chronic Intake of Cannabis on Contrast Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5331; 2012-A00991-42 (Other: n° IDRCB)
Record Dates: First submitted 2013-02-12; First posted 2013-02-18 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Cannabis Dependence
MeSH Terms: conditions — Marijuana Abuse

ARMS (3):
- "Cannabis" Arm (Other): patient addicted to cannabis
  Interventions: Other: electroretinogram; Other: contrast sensitivity tests
- "Tobacco" Arm (Other): patient addicted to tobacco
  Interventions: Other: electroretinogram; Other: contrast sensitivity tests
- "Healthy volunteers" (Other): no smokers
  Interventions: Other: electroretinogram; Other: contrast sensitivity tests

INTERVENTIONS:
Other: electroretinogram
Other: contrast sensitivity tests

SUMMARY:
Rates of driving under the influence of cannabis have risen in recent years. Cannabis is involved in 1/3 of motor vehicle collisions. The chronic use of cannabis is known to affect dopaminergic regulation and may thus impair contrast sensitivity. In turn, contrast sensitivity disorders could originate difficulties to anticipate and avoid collision with objects, especially when objects are in movement. The investigators goal is to examine the effects of a chronic intake of cannabis on contrast sensitivity. The observed values will be compared to standard references. In addition, since smoking cannabis is always associated with tobacco, the investigators will control the effects of tobacco on contrast sensitivity.

In this study, the investigators will include 36 cannabis addicts, 36 tobacco addicts and 36 no smokers. The investigators will present gratings with different spatial frequencies and the investigators will determine contrast thresholds for static and dynamic (moving) gratings. The investigators predict that cannabis addicts will present abnormal contrast sensitivity especially in case of dynamic presentation of gradings.

ELIGIBILITY:
Inclusion Criteria:

"Cannabis" Arm

* patient addicted to cannabis
* Positive CAST test result
* Urine tested positive for cannabis metabolites

"Tobacco" Arm

* positive Fagerström test result
* No cannabis intake in the last year before inclusion
* No previous history of cannabis use

"Healthy Volunteers"

* No tobacco or cannabis intake in the last year before inclusion
* No history of addictive disorders

Exclusion Criteria:

* addiction to other substances than cannabis or tobacco
* benzodiazepine treatment
* patient with history of benzodiazepine treatment
* patient with history of general anesthesia in the last 3 months before inclusion
* patient with history of head trauma
* Pregnant woman
* breast feeding woman
* Adults under supervision or guardianship

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2013-03-22 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
The contrast detection treshold | up to 9 days after inclusion
  Comparison of the contrast detection threshold of the 3 groups